CLINICAL TRIAL: NCT01784653
Title: Randomized Controlled Trial of Computerized MET for Adolescent Substance Use
Brief Title: Trial of Computerized MET for Adolescent Substance Use
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No funding obtained.
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Sion Kim Harris, Co-Director, Center for Adolescent Substance Abuse Research, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKH R01 PA-13-077
Record Dates: First submitted 2013-02-04; First posted 2013-02-06 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Drug Abuse; Alcohol Abuse; Nicotine Dependence
Keywords: Substance abuse; Drug abuse; Alcohol abuse; Tobacco; Adolescent
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism; Tobacco Use Disorder | interventions — histaminol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment as Usual (No Intervention): Patients will receive the usual care from the treatment program
- iMET (Experimental): Participants will complete a self-guided computerized Motivational Enhancement Therapy
  Interventions: Behavioral: iMET
- MET (Experimental): Clinician-delivered Motivational Enhancement Therapy
  Interventions: Behavioral: MET

INTERVENTIONS:
Behavioral: iMET — Self-completed, computerized motivational enhancement therapy
  Arms: iMET
Behavioral: MET — Clinician-delivered Motivational Enhancement Therapy
  Arms: MET

SUMMARY:
The purpose of this study is to test the effects of a computerized, self-directed Motivational Enhancement Therapy program for adolescent substance use (iMET), in comparison to clinician-delivered MET and Treatment As Usual (TAU), on treatment engagement and substance use. The investigators hypothesize that both iMET and MET will be more effective than TAU in engaging/retaining patients in treatment and in reducing substance use during a 12-month follow-up period. The investigators also hypothesize that Self-directed iMET will be as effective as the clinician-guided MET in increasing treatment engagement and abstinence during the 12-months follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* completed initial visit at the treatment program;
* be available to return for iMET/MET sessions (if assigned)
* be available to complete all follow-up measurements
* a past-12-month CRAFFT score >1
* have used substances on >6 days (not including tobacco use) during the 90 days preceding their visit

Exclusion Criteria:

* unable to speak and understand English, or read English at a 5th grade reading level
* youth deemed by the clinical team to require immediate hospitalization or referral to more intensive residential treatment

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Treatment engagement | 12 months
  We will compare the number of individual visits in the program, the number of group sessions completed, and the number of urine screens completed during a 12 month follow-up period by each participant in the three study arms.

SECONDARY OUTCOMES:
Days abstinent | past-90-days
  We will calculate the past-90-days number of days abstinent from any substance use and from the primary substance and the number of weeks abstinent from any substance use.
Driving/Riding Risk | past-90-days
  We will compare group trends in prevalence and frequency of past-90-days Driving while impaired or Riding with an impaired driver.
HIV Risk Behavior | past-90-days
  We will compare group trends in prevalence and frequency of past-90-days HIV Risk Behaviors.

OTHER OUTCOMES:
Treatment process/quality | 60 days
  We will compare completion of the 2 MET sessions, and completion of the third follow-up visit between the iMET and MET conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Sion K Harris, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States